CLINICAL TRIAL: NCT06234683
Title: Assessing Barriers to Pneumococcal Vaccination to Increase Vaccine Uptake Among Older Adults: a Web-based Educational Intervention
Brief Title: PRomoting Older Adults' Pneumococcal Vaccination Through Education and Learning
Acronym: PROPEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CIRN Project SH-34
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-04

CONDITIONS: Pneumococcal Vaccine Uptake; Vaccination Willingness; Pneumococcal Vaccine Knowledge; Pneumococcal Vaccine Attitude
Keywords: pneumococcal vaccines; older adults; vaccine hesitancy; health education; web-based intervention
MeSH Terms: conditions — Vaccination Hesitancy; Health Education

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to receive either a web-based educational video about pneumococcal vaccination and a reminder email to be vaccinated or a reminder email alone.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Web-based educational video on pneumococcal vaccination and reminder email to be vaccinated (Active Comparator)
  Interventions: Other: Web-based educational video on pneumococcal vaccination; Other: Reminder email to be vaccinated
- Reminder email to be vaccinated (Placebo Comparator)
  Interventions: Other: Reminder email to be vaccinated

INTERVENTIONS:
Other: Web-based educational video on pneumococcal vaccination — Participants will receive a link to view a short video on pneumococcal vaccination.
  Arms: Web-based educational video on pneumococcal vaccination and reminder email to be vaccinated
Other: Reminder email to be vaccinated — Participants will receive a reminder email to be vaccinated.

SUMMARY:
The goal of this trial is to compare the effect of a web-based educational video about pneumococcal vaccines and a reminder email to get vaccinated (intervention) with a reminder email alone (comparator) in adults aged 65 or older living in any Canadian province who reported not having received a pneumococcal vaccine.

The main questions this trial aims to answer are:

1. does the educational intervention improve pneumococcal vaccine uptake,
2. does the educational intervention improve willingness to be vaccinated,
3. does the educational intervention improve knowledge of pneumococcal vaccination,
4. and does the educational intervention improve attitudes towards pneumococcal vaccines/vaccination?

Eligible participants who provide electronic consent will:

1. fill out a web-based baseline survey,
2. receive access to the educational video (if assigned to the intervention group),
3. receive an email reminder to be vaccinated (both groups),
4. and fill in a web-based follow-up survey.

DETAILED DESCRIPTION:
This research project is a web-based randomized controlled trial (RCT), targeting adults aged 65 years and older across all Canadian provinces. The primary objectives of this study are twofold. Firstly, it aims to assess the participants' knowledge, barriers, facilitators, and willingness to receive the pneumococcal vaccine at baseline. Secondly, it aims to evaluate the impact of a video-led educational intervention on pneumococcal vaccine literacy, willingness to be vaccinated, and the actual uptake of the vaccine. To this end, participants will be recruited through various online channels. Only individuals who have not received the pneumococcal vaccine will be considered eligible for inclusion. For the second objective, participants will be randomly assigned to either the intervention group (short video on pneumococcal vaccination) or the control group (reminder to receive a pneumococcal vaccine). Consenting participants will be required to complete two surveys: one at baseline and another approximately six months post-intervention. These surveys will provide valuable data for analyzing the effectiveness of the educational intervention in improving participants' knowledge, willingness to be vaccinated, and the actual uptake of the pneumococcal vaccine. Findings from this research will contribute to the understanding of factors influencing pneumococcal vaccine decision-making among older adults, ultimately informing strategies to enhance vaccine uptake and public health outcomes in this population.

ELIGIBILITY:
Inclusion criteria:

1. adults aged ≥ 65 residing in any Canadian province,
2. community dwelling (i.e., living outside of nursing homes),
3. reporting not having received a pneumococcal vaccine, and
4. being able to understand English and/or French.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 720 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Pneumococcal vaccine uptake measured using a web-based follow-up survey four to six months post-randomization | 4-6 months
  Participants will be asked at follow-up whether they received a pneumococcal vaccine since the last survey (yes/no/do not know).

SECONDARY OUTCOMES:
Change in pneumococcal vaccination willingness, measured using web-based surveys (one at baseline and one four to six months post-randomization) | 4-6 months
  Participants will be asked at baseline and follow-up whether they would be willing to receive a pneumococcal vaccine (yes/no/do not know).
Change in pneumococcal vaccine knowledge measured using web-based surveys (one at baseline and one four to six months post-randomization) | 4-6 months
  Participants will be asked about their vaccine knowledge at baseline and follow-up (yes/no/do not know).
Change in pneumococcal vaccine attitudes measured using web-based surveys (one at baseline and one four to six months post-randomization) | 4-6 months
  Participants will be asked about their vaccine attitudes using Likert-type questions at baseline and follow-up. The response options are on a 5-point Likert scale that ranges from a value of 1 for strongly disagree to a value of 5 for strongly agree. Higher scores indicate stronger agreement with the statement and with the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgia Sulis, PhD, Principal Investigator — School of Epidemiology and Public Health, Faculty of Medicine, University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No